CLINICAL TRIAL: NCT00005911
Title: Refinement of the Magnetic Resonance Imaging Technique for the Study of the Normal Eye, Particularly the Lens and Cataract
Brief Title: Magnetic Resonance Imaging to Study the Normal Eye
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000151; 00-EI-0151
Record Dates: First submitted 2000-06-13; First posted 2000-06-14 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-08

CONDITIONS: Cataract; Lens Disease
Keywords: Magnetic Resonance Imaging; Human Eye; Lens; Normal Volunteers; Cataract; Human Lens; Healthy Volunteer
MeSH Terms: conditions — Cataract; Lens Diseases

SUMMARY:
This study will assess the value of improved magnetic resonance imaging (MRI) techniques to study the lens of the human eye. Knowledge of how cataracts develop and progress has been hampered by the lack of human tissue available for study; MRI may provide an effective means for learning more about this eye disease.

Normal volunteers between 18 and 70 years of age may be eligible for this study. Participants will undergo a medical history and complete eye examination, including vision assessment, eye pressure measurement, lens and retina examinations, and photography of the eye.

MRI scans will be scheduled for a second visit. For this procedure, the volunteer's pupils are dilated and he or she then lies on a stretcher that is moved into a cylinder containing a magnetic field. A device similar to a welder's helmet is placed on the head. Attached to the device are an imaging probe and a small blinking light. The probe receives radio signals from the eye that a computer converts into images. During imaging, the participant gazes at the blinking light; this helps keep the eyes from blinking and wandering. Scan times vary from 2 to 10 minutes; the total time for the study is less than an hour.

DETAILED DESCRIPTION:
Studies of human diabetic cataract and age related cataract formation have been hampered by unavailability of human tissues especially in the early stages of the disease. Eye bank tissues are first used for cornea transplants so that by the time they become available for basic research studies, the lens is no longer suitable for biochemical nor histological studies. Cataracts usually only become available after extraction which is at the end stage of their development. However, appropriate surgical lens specimens are no longer available because cataracts are generally extracted by the destructive phakoemulsification technique. Therefore, noninvasive techniques are required in order to study the lens in vivo.

ELIGIBILITY:
Must be between 18 and 70 years of age of either sex.

Must not have uveitis, glaucoma, or be at risk for an adverse reaction to dilation or have a history of allergic reaction to one of lthe dilating agents to be used.

Must not have any metallic prosthesis, cardiac pacemakers, neural pacemakers, surgical clips in the brain or on blood vessels, surgically implanted metal plates, screws or pins, cochlear implants or metal objects in the body especially in the eye.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 2000-06; Study Completion 2002-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Kinoshita JH, Kador P, Catiles M. Aldose reductase in diabetic cataracts. JAMA. 1981 Jul 17;246(3):257-61. No abstract available. PMID 6787220
- [Background] Reddy VN, Schwass D, Chakrapani B, Lim CP. Biochemical changes associated with the development and reversal of galactose cataracts. Exp Eye Res. 1976 Nov;23(5):483-93. doi: 10.1016/0014-4835(76)90157-3. No abstract available. PMID 1001376
- [Background] Datiles M, Fukui H, Kuwabara T, Kinoshita JH. Galactose cataract prevention with sorbinil, an aldose reductase inhibitor: a light microscopic study. Invest Ophthalmol Vis Sci. 1982 Feb;22(2):174-9. PMID 6799419